CLINICAL TRIAL: NCT01960088
Title: Building Evidence to Expand Adolescent Vaccination in Pharmacies
Brief Title: Adolescent Vaccination in Pharmacies
Acronym: AVIP
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-2889
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Evaluating Attitudes Toward HPV Vaccinations in Pharmacies; Evaluating the Provision of HPV Vaccines in a Pharmacy
Keywords: Adolescent vaccines; HPV vaccine; Pharmacies
MeSH Terms: interventions — Papillomavirus Vaccines; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — N=1200 anticipated in national study N=100 anticipated in pharmacy demonstration project
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adolescents and their parents: Pharmacy demonstration project: HPV vaccine delivery
  Interventions: Drug: HPV vaccine

INTERVENTIONS:
Drug: HPV vaccine
  Other Names: Gardasil

SUMMARY:
The study aims to expand the evidence supporting pharmacy provision of adolescent vaccines, including human papillomavirus (HPV) vaccine. In the first part of the study, we will characterize parents' attitudes and support for pharmacy provision of adolescent vaccines in a national survey. In the second part of the study, we will provide HPV vaccines and other vaccines (Tdap, meningococcal, varicella, influenza) to 200 adolescents in a local community pharmacy in Chapel Hill, North Carolina. This portion of the study will identify the systems and workflow needed to provide vaccines effectively and safely, characterize parents' and their adolescents' attitudes toward receiving vaccine services in a pharmacy, and characterize pharmacists' attitudes toward providing adolescent vaccine services in a pharmacy.

ELIGIBILITY:
NATIONAL SURVEY (probability sample)

Inclusion Criteria:

* Being a member of the GfK Knowledge Panel
* Having a child age 11-18.

Exclusion Criteria:

● None

PHARMACY DEMONSTRATION PROJECT (convenience sample)

Inclusion Criteria:

* Having an adolescent child, ages 11-18 years old, who is healthy, and for whom HPV vaccine is indicated
* Child is with the parent

Exclusion Criteria:

● Being the parent of an adolescent who is immunocompromised, or has other chronic illness, has known anaphylactoid/hypersensitivity reactions to components of HPV vaccine used, or is pregnant or plan to be pregnant within a month of vaccination.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: National survey: Parents of adolescents ages 11-18. Pharmacy sample: Parents of adolescent boys and girls, ages 11-18 whose families reside in the Chapel Hill area, and their adolescents.
Sampling Method: Non-Probability Sample
Enrollment: 1509 (Actual)
Dates: Start 2015-07; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Parents' willingness to get their adolescent children HPV vaccine in pharmacy | At time of study
  Outcome is for the national survey of parents.
Parents' satisfaction with HPV vaccine vaccine administration in the pharmacy | At time of vaccine administration
  Outcome is for demonstration study in a community pharmacy.

CONTACTS AND LOCATIONS:
Overall Officials: Noel T Brewer, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Central Pharmacy, Durham, North Carolina
  - Triangle Pharmacy, Durham, North Carolina